CLINICAL TRIAL: NCT04026230
Title: Impact of Atorvastatin on Prostate Cancer Progression After Initiation of Androgen Deprivation Therapy - Lipid Metabolism as a Novel Biomarker to Predict Prostate Cancer Progression
Brief Title: Impact of Atorvastatin on Prostate Cancer Progression During ADT
Acronym: ESTO2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Central Finland Hospital District (Other); Tartu University Hospital (Other); University of Aarhus (Other); Fimlab laboratories (Unknown); Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Seinajoki Central Hospital (Other); The Hospital of Vestfold (Other); Telemark Hospital Trust (Unknown)
Responsible Party: Principal Investigator, Teemu Murtola, MD, PhD, professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-004774-17
Record Dates: First submitted 2018-06-25; First posted 2019-07-19 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Prostate Cancer; Recurrent Prostate Cancer
Keywords: Prostate cancer; Castration resistance; Cholesterol lowering drug; Cholesterol; Atorvastatin; Survival; Mortality
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Experimental): Capsules of atorvastatin. Daily dose of 80 mg for max. 10 years or until development of castration resistance.
  Interventions: Drug: Atorvastatin 80mg
- Placebo (Placebo Comparator): Identical capsules as in the atorvastatin arm, but including no active ingredient. Used daily for max. 10 years or until development of castration resistance
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Atorvastatin 80mg — Capsules including 80 mg of atorvastatin
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo oral capsule — Similar capsules as in the atorvastatin arm, but without the active ingredient
  Arms: Placebo

SUMMARY:
This randomized double-blind placebo-controlled trial tests whether intervention with atorvastatin delays development of castration resistance compared to placebo during androgen deprivation therapy (ADT) for prostate cancer.

DETAILED DESCRIPTION:
Cholesterol-lowering statin drugs have been reported to lower proliferation activity in prostate cancer, delay occurrence of castration resistance and reduce the risk of prostate cancer death. Therefore, it is important to test statins' efficacy in addition to conventional prostate cancer treatment in a randomized, placebo-controlled trial.

This phase 3 randomized double-blind placebo-controlled trial will explore whether intervention with atorvastatin delays prostate cancer progression i.e. development of castration resistance compared to placebo during androgen deprivation therapy (ADT) for metastatic or recurrent prostate cancer.

Secondary objectives include exploring whether atorvastatin lowers prostate cancer-specific or overall mortality compared to placebo, and to demonstrate whether changes in serum lipid parameters predict disease recurrence and occurrence of adverse genomic changes predicting castration resistance among prostate cancer patients during ADT.

The study recruitment target is 400 participants who start ADT as management of metastatic or recurrent prostate cancer. These men will be randomized 1:1 (200 + 200) to receive blinded study drug, either 80 mg of atorvastatin daily or placebo until disease recurrence i.e. development of castration resistance or for a maximum of five years.

The study will be carried out in collaboration between urological departments of University Hospitals in Finland as a project of the national FinnProstata study group, Herlev University Hospital in Denmark, Vestfold and Telemark hospitals in Norway and the Tartu University Hospital in Estonia.

Follow-up is continued until the primary end-point, development of castration resistance. After this the participants will be given the opportunity to voluntarily carry on with the blinded intervention for maximum time of ten year to observe effects on survival after development of castration resistance. Blinding will be lifted after the follow-up is complete for all study participants.

Castration resistance is defined as prostate-specific antigen (PSA) progression (three consecutive rises of PSA measured at least 1 week apart with two > 50% increases over the nadir and PSA > 2 ng/ml) or radiological disease progression (appearance of two or more lesions in bone scan or soft tissue enlargement as per RECIST criteria) with serum testosterone at castrate level (< 1.73 nmol/l; 50 ng/dl) during ADT.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed metastatic (radiologically confirmed bone or soft tissue metastasis or enlarged lymph nodes at minimum 15 mm in diameter beyond the pelvic lymph nodes) or recurrent (requiring treatment after curative-intent surgery or radiotherapy) adenocarcinoma of the prostate for which androgen deprivation or antiandrogen therapy (GnRH agonist/antagonist, bicalutamide/flutamide, surgical castration or enzalutamide/abiraterone monotherapy) is initiated as definitive treatment no longer than 3 months before recruitment

  * previous prostatectomy and radiation therapy allowed
  * ADT/antiandrogen therapy for neoadjuvant hormone therapy is not included
* Willingness to participate and signing of informed consent

Exclusion Criteria:

* Statin use at the time of recruitment or within 6 months of it
* Previous adverse effects during statin therapy
* Familial hypercholesterolemia or very high total cholesterol (9.3 mmol/l or above)
* Clinically significant renal insufficiency (serum creatinine above 170 µmol/l) or liver insufficiency (serum alanine aminotransferase more than 2x above the upper limit of normal range)
* Use of drugs that may interact with statins (St John's Wort, HIV protease inhibitors, ciclosporin, macrolide antibiotics, fucidic acid, phenytoin, carbamazepine, dronedarone or oral antifungal medication).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Castration resistance | From date of randomization until the date of first occurrence of castration resistance, assessed up to 60 months
  Castration resistance is defined as PSA progression (three consecutive PSA rises measured at least 1 week apart with two > 50% increases over the nadir and PSA > 2 ng/ml) or radiological disease progression (appearance of two or more lesions in bone scan or soft tissue enlargement as per RECIST criteria) with serum testosterone at castrate level (< 1.73 nmol/l; 50 ng/dl) during ADT.

SECONDARY OUTCOMES:
Lipid levels | From date of randomization until the date of first occurrence of castration resistance or death, whichever came first, assessed at 6 month intervals up to 60 months
  Change in serum lipid levels during the intervention. Measured at baseline and in every follow-up visit. Results are blinded from the investigators and participants before the final analysis
Prostate cancer mortality | From date of randomization until the date of prostate cancer death, assessed up to 60 months
  Followed through Finnish national registries after reaching the primary end-point
Overall survival | From date of randomization until the date of death due to any cause, assessed up to 60 months
  Followed through Finnish national registries after reaching the primary end-point
Circulating cell-free DNA | At enrollment and at occurrence of castration resistance, assessed up to 60 months
  Occurrence of adverse tumor traits predicting development of castration resistance in circulating cell free DNA
Fasting blood glucose | From date of randomization until the date of first occurrence of castration resistance or death, whichever came first, assessed at 6 month intervals up to 60 months
  To see how ADT affects glucose tolerance and whether atorvastatin intervention has any effect on it
Occurrence of cardiovascular events during ADT | From date of randomization until the date of first occurrence of castration resistance or death, whichever came first, assessed at 6 month intervals up to 60 months
  Any cardiovascular events as described by the participant or evident from the patient files during the course of follow-up. Followed via national registries after meeting the primary end-point.
General quality of life (QOL) | From date of randomization until the date of first occurrence of castration resistance or death, whichever came first, assessed at 12 month intervals up to 60 months
  Score from validated QOL questionnaire EORTC QLQ-C30 (range 0-100, with 100 denoting highest quality of life)
Prostate cancer-specific quality of life (QOL) | From date of randomization until the date of first occurrence of castration resistance or death, whichever came first, assessed at 12 month intervals up to 60 months
  Score from validated QOL questionnaire EORTC QLQ-PR25 (range 0-100, with 100 denoting highest quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Murtola, MD, PhD, Principal Investigator — Tampere University Hospital; Otto Ettala, MD, PhD, Study Director — Turku University Hospital; Heikki Seikkula, Study Director — Central Finland Central Hospital
Locations (10):
- Herlev and Gentofte Hospital, Herlev, Denmark
- Tartu University Hospital, Tartu, Estonia
- Finland (6):
  - Helsinki University Hospital, Department of Urology, Helsinki
  - Central Finland central hospital, Jyväskylä
  - Kuopio University Hospital, Department of Urology, Kuopio
  - Seinäjoki Central Hospital, Department of Surgery, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Norway (2):
  - The Hospital of Telemark, Skien
  - The Hospital of Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: No
Sharing of individual-level data is not allowed by ethics board

REFERENCES:
- [Derived] Siltari A, Riikonen J, Koskimaki J, Pakarainen T, Ettala O, Bostrom P, Seikkula H, Kotsar A, Tammela T, Helminen M, Raittinen PV, Lehtimaki T, Fode M, Ostergren P, Borre M, Rannikko A, Marttila T, Salonen A, Ronkainen H, Loffeler S, Murtola TJ. Randomised double-blind phase 3 clinical study testing impact of atorvastatin on prostate cancer progression after initiation of androgen deprivation therapy: study protocol. BMJ Open. 2022 Apr 29;12(4):e050264. doi: 10.1136/bmjopen-2021-050264. PMID 35487730